CLINICAL TRIAL: NCT03938974
Title: The Emergence and Evolution of Social Self-Management of Parkinson's Disease
Brief Title: Social Self-Management of Parkinson's Disease
Acronym: SocM-PD
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Linda Tickle-Degnen, Professor, Tufts University
Other Study IDs: 1212038; R01NR013522 (NIH)
Record Dates: First submitted 2019-04-17; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Parkinson Disease
Keywords: self-management; social ecology; biopsychosocial; social participation; everyday living; person-centered; longitudinal
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parkinson's disease (PD) affects 1% to 2% of the US population over age 60, and its prevalence is increasing as the population ages. The proposed research will establish the natural evolution of the social lives of people with Parkinson's disease and their families and its relationship to health outcomes, and thus has the potential to significantly advance Parkinson's disease research and evidence-based neurological nursing and rehabilitation. The project develops the new construct of social self-management of chronic disease and results will inform the development of new interventions aimed at supporting social integration and preventing isolation and loneliness in people living with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD), one of the most common age-related neurodegenerative disorders, affects facial, vocal and trunk muscles. As this progressive decline occurs, an expressive mask descends, limiting the person's ability to communicate emotions and intentions to others, which may give the impression that the person is cold, asocial or apathetic. Thus, as people with PD are living longer and residing in their homes longer, the burden of care-giving is unmitigated by the social and emotional rewards provided by an expressive individual. While this disability has been discussed in the literature, relatively little is known about how adults living with a chronic physical disease such as PD manage their social lives and how an inability to be emotionally expressive can affect social connections. Because social networks have been shown to be crucial to the overall well-being of people living with chronic diseases, research on how expressive capacity affects life trajectories and overall health is critically needed. The overall objective of this project is to understand the emergence and evolution of social self-management trajectories of people living with PD, and this work has the potential to significantly advance PD research and evidence-based neurological nursing and rehabilitation. The investigators will test the central hypothesis that PD expressive capacity predicts systematic change in the pattern of social self-management of PD and quality of life outcomes.

The Specific Aims of this three-year longitudinal study of 120 patients with PD and a maximum of 120 care partners are: 1) Characterize social self-management trajectories of individuals with PD over a three-year period; 2) Estimate the degree to which expressive nonverbal capacity predicts the social self-management trajectory; and 3) Determine the moderating effect of gender on the association between expressive capacity and change in social self-management.

Over the three-year project period, investigators will assess patients with PD and a care partner 14 times each to examine such factors as social participation and management of social activities; social network; and social comfort, general health and well-being. Descriptive analyses will be performed on the total sample and on meaningful demographic and clinical subgroups. This study is designed to have sufficient power to detect changes over time and to detect differences in gender. The investigators' contribution is significant because it will provide evidence to guide the development of interventions aimed at supporting social integration of people living with PD, thus leading to improved overall health. The proposed work is innovative because, to the best of the investigators' knowledge, it is the first to focus on the novel construct of social self-management and does so in a manner that reflects the daily lived experience of PD. Further, the investigators go beyond descriptive evidence to rigorously test hypotheses regarding factors known to contribute to social stigmatization, expressive capacity and gender.

ELIGIBILITY:
Inclusion Criteria for People with Parkinson's Disease:

1. Diagnosis of idiopathic PD utilizing the UK Parkinson's Disease Society Brain Bank clinical diagnostic criteria, as evaluated by the neurological team
2. Modified Hoehn and Yahr stage 1 through 4
3. Score ≥ 26 on the Mini-Mental Status Exam
4. Home setting within travel distance to study locations
5. Able to communicate clearly and in English with research staff
6. Interested in participating and willing and able to provide informed consent

Inclusion Criteria for Care Partners of Participants with Parkinson's Disease:

1. Person with PD must consent for care partner to participate
2. Score ≥ 26 on the Mini-Mental Status Exam
3. Able to communicate clearly and in English with research staff
4. Interested in participating and willing and able to provide informed consent

Exclusion Criteria for People with Parkinson's Disease:

1. Diagnosis of atypical Parkinsonism
2. Modified Hoehn and Yahr Stage 5
3. Score < 26 on the Mini-Mental Status Exam
4. Not able to communicate clearly and in English with research staff

Exclusion Criteria for Care Partners of Participants with Parkinson's Disease:

1. Person with PD does not consent for care partner to participate
2. Score < 26 on the Mini-Mental Status Exam
3. Not able to communicate clearly and in English with research staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We recruited People with Parkinson's disease as primary participants (Care partners were enrolled if available) through the Boston University Medical Center Parkinson's Disease and Movement Disorders Clinic, regional Parkinson's disease support groups, older adult service centers, and postings on research and advocacy websites. The neurological medical team conducted and supervised the medical history and screening.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2013-09-23 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Activity Retention Over Time | 3 Years
  Activity Card Sort domains of Instrumental Activities of Daily Living, Low- and High-Demand Leisure Activities, and Social Activities.
The Chronic Illness Resources Survey (CIRS) | 3 Years
  The 22-item CIRS, slightly modified for this study. Respondents rate the extent to which each of the 22 items is accessible or used as a resource over the past 6 months on a 1 (not at all) to 5 (a great deal) Likert scale. Subscale scores are created by averaging (possible range 1 to 5), and include the following: Personal Self-Management (3 items); formal institutions and services-- Health Care (3 items), Organizations (3 items), Work (3 items) and Media and Policy (3 items); and informal interpersonal environment-- Family and Friends (3 items) and Neighborhood (3 items). CIRS was modified by changing the wording of "chronic illness" to "health management." Higher scores represent a better outcome (i.e., greater access to and utilization of healthy resources).
Social Network Composition | 3 Years
  Self-reported responses to the following items: having a spouse or partner in the household (yes/no), number and composition of individuals living in the household, total number of children and total number of grandchildren.
Contact Frequency | 3 years
  How often, on a 0 (not at all) to 7 (very frequently), are participants in contact with the following:
  Their most contacted child (if they have children) Their most contacted friend (if they have friends) Their partner in the study (if applicable)
Support Exchange | 3 Years
  Rated on a scale from 1 (not at all) to 5 (a great deal), how often do participants give different types of support (Help with Daily Activities, Emotional Support, and Financial Support) to either their partner in the study (if applicable), the members of their household, and people outside of their household.
Social Isolation Domain of the Nottingham Health Profile (NHP) | 3 Years
  The Social Isolation Domain of the NHP is a 5-item measure: loneliness, difficulty contacting people, feeling that they have no one they are close to, difficulty getting along with others, and feeling like a burden. Participants rate their agreement with statements related to social isolation on a scale from 1 (extremely disagree) to 5 (highly agree) and these items are averaged. A higher score is a worse outcome.
The Positive Social Interaction subscale items of the Medical Outcomes Study: Social Support Survey (MOS) | 3 Years
  We modified the wording of the three Positive Social Interaction items in the MOS Social Support Survey to identify positive interaction frequency with the care partner or the person with PD, rather than a non-specific "someone." Our wording is: "How often is each of the following kinds of support available to you from your partner if you need it?" Each item is rated on a 1 (None of the time) to 5 (All of the time) scale, and these items are averaged. A higher score indicates a better outcome.
The Stigma Scale for Chronic Illness (SSCI) | 3 Years
  The 24-item SSCI has two domains: felt stigma and enacted stigma. Felt stigma items assess the emotional experience of stigmatization such as worry, embarrassment and self-blaming. Enacted stigma items assess the perception that people act differently toward the respondent: acting uncomfortable, being unkind, avoiding contact, and unfair treatment. Each domain contains 12 items (which are averaged to create domain scores), rated on a scale from 1 (never) to 5 (always). A total score is calculated by averaging all items. A higher score is a worse outcome and indicates greater stigma.
The Interpersonal Communication Rating Protocol: Individual Expressive Behavior (Parkinson's Disease Version) (ICRP-IEB) | 3 Years
  The 20-item ICRP-IEB is used as the primary measure of the expressive capacity of participants with PD coded from videotaped discussions. Four to ten trained coders rate the videos on a scale from 1 (low) to 5 (high) of the intensity, duration, and frequency of expressive behaviors from the following domains: facial, bodily, vocal, and verbal. Scores are averaged within domains. A higher score is a better outcome and indicates more expressive behaviors.
Qualitative Self-Management Interview | 3 Years
  Self-identified frustrating and satisfying recent events in daily life and how they manage these and similar events. Next, participants describe an activity outside of the home and how they get ready for it and manage PD symptoms to do it. Finally, participants are asked - How would you rate your overall ability to manage participating in your daily life activities? They provide a response on a scale of 1 (not at all effective) to 5 (highly effective). Participants with PD are videotaped and care partners are audiotaped.
  In a second management discussion, we bring together the person with PD and the caregiver and ask them to think of an activity outside of the home that they recently did together. The discussion is videotaped with the camera focused only on the participant with PD.
  One of the interviews is conducted in participants' homes, midway through the three-year protocol.

SECONDARY OUTCOMES:
Short Form -12 (SF-12, version 2) | 3 Years
  The 12-item SF-12 (version 2) is a self-report measure of functional health and well-being that is a short form of the SF-36. It provides norm-based scores in two domains (physical and mental health), that compare the respondent against population level health. A higher score is better outcome for health.
The Parkinson's Disease Questionnaire-39 (PDQ-39) | 3 years
  The PDQ-39 assesses life concerns of individuals with PD. It is composed of a summary index and eight domain scores-mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and bodily discomfort. Each item is rated on a 0 (never) to 4 (always) scale. A higher score indicates a higher self-perceived frequency of quality of life and health problems in the past month that are due to the disease, with each domain normed to a scale on which 0 indicating never a problem and 100 always a problem. The summary index is the average of the normed domain scores. A higher score is a worse outcome for quality of life.
The Movement Disorder Society Unified Parkinson's Disease Rating Scales (MDS-UPDRS). | 3 Years
  The Movement Disorder Society's Unified Parkinson's Disease Rating Scales (MDS-UPDRS) consists of 65 items across four domains: non-motor experiences, motor experiences, a motor examination, and motor complications, rated from 0 (normal) to 4 (severe). Subscales and a total score are calculated by adding items. A higher score is worse outcome and indicates more severe symptoms of Parkinson's disease.
The Geriatric Depression Scale-15 (GDS) | 3 Years
  The GDS consists of 15 yes or no items. The total score is the sum of all items (range: 0 - 15). A higher score is a worse outcome and indicates greater potential for clinical depression.
The Montreal Cognitive Assessment (MoCA) | 3 Years
  The MoCA consists of 30 test items that assess visuospatial and executive functioning, naming, memory, attention, language, abstraction, delayed recall, and orientation. Each correct answer is awarded one point, which are added to create a total score. A higher score is a better outcome and indicates less cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Tickle-Degnen, PhD, Principal Investigator — Tufts University
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Tufts University, Medford, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alves G, Wentzel-Larsen T, Aarsland D, Larsen JP. Progression of motor impairment and disability in Parkinson disease: a population-based study. Neurology. 2005 Nov 8;65(9):1436-41. doi: 10.1212/01.wnl.0000183359.50822.f2. PMID 16275832
- [Background] Ambady N, Koo J, Rosenthal R, Winograd CH. Physical therapists' nonverbal communication predicts geriatric patients' health outcomes. Psychol Aging. 2002 Sep;17(3):443-452. doi: 10.1037/0882-7974.17.3.443. PMID 12243386
- [Background] Ambady N, Laplante D, Nguyen T, Rosenthal R, Chaumeton N, Levinson W. Surgeons' tone of voice: a clue to malpractice history. Surgery. 2002 Jul;132(1):5-9. doi: 10.1067/msy.2002.124733. PMID 12110787
- [Background] Bogart KR. Is apathy a valid and meaningful symptom or syndrome in Parkinson's disease? A critical review. Health Psychol. 2011 Jul;30(4):386-400. doi: 10.1037/a0022851. PMID 21480712
- [Background] Bogart KR, Tickle-Degnen L, Ambady N. Compensatory expressive behavior for facial paralysis: adaptation to congenital or acquired disability. Rehabil Psychol. 2012 Feb;57(1):43-51. doi: 10.1037/a0026904. PMID 22369116
- [Background] Bogart KR, Tickle-Degnen L, Joffe MS. Social interaction experiences of adults with Moebius Syndrome: a focus group. J Health Psychol. 2012 Nov;17(8):1212-22. doi: 10.1177/1359105311432491. Epub 2012 Jan 18. PMID 22257565
- [Background] Buchman AS, Boyle PA, Wilson RS, Fleischman DA, Leurgans S, Bennett DA. Association between late-life social activity and motor decline in older adults. Arch Intern Med. 2009 Jun 22;169(12):1139-46. doi: 10.1001/archinternmed.2009.135. PMID 19546415
- [Background] Buchman AS, Boyle PA, Wilson RS, James BD, Leurgans SE, Arnold SE, Bennett DA. Loneliness and the rate of motor decline in old age: the Rush Memory and Aging Project, a community-based cohort study. BMC Geriatr. 2010 Oct 22;10:77. doi: 10.1186/1471-2318-10-77. PMID 20969786
- [Background] Chastin SF, Baker K, Jones D, Burn D, Granat MH, Rochester L. The pattern of habitual sedentary behavior is different in advanced Parkinson's disease. Mov Disord. 2010 Oct 15;25(13):2114-20. doi: 10.1002/mds.23146. PMID 20721926
- [Background] Dahodwala N, Siderowf A, Xie M, Noll E, Stern M, Mandell DS. Racial differences in the diagnosis of Parkinson's disease. Mov Disord. 2009 Jun 15;24(8):1200-5. doi: 10.1002/mds.22557. PMID 19412929
- [Background] Davis LL, Weaver M, Habermann B. Differential attrition in a caregiver skill training trial. Res Nurs Health. 2006 Oct;29(5):498-506. doi: 10.1002/nur.20138. PMID 16977645
- [Background] Duncan RP, Earhart GM. Measuring participation in individuals with Parkinson disease: relationships with disease severity, quality of life, and mobility. Disabil Rehabil. 2011;33(15-16):1440-6. doi: 10.3109/09638288.2010.533245. Epub 2010 Nov 20. PMID 21091047
- [Background] Eagly AH. The his and hers of prosocial behavior: an examination of the social psychology of gender. Am Psychol. 2009 Nov;64(8):644-58. doi: 10.1037/0003-066X.64.8.644. PMID 19899859
- [Background] Everard KM, Lach HW, Fisher EB, Baum MC. Relationship of activity and social support to the functional health of older adults. J Gerontol B Psychol Sci Soc Sci. 2000 Jul;55(4):S208-12. doi: 10.1093/geronb/55.4.s208. PMID 11584883
- [Background] Forsaa EB, Larsen JP, Wentzel-Larsen T, Herlofson K, Alves G. Predictors and course of health-related quality of life in Parkinson's disease. Mov Disord. 2008 Jul 30;23(10):1420-7. doi: 10.1002/mds.22121. PMID 18512757
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Glasgow RE, Strycker LA, Toobert DJ, Eakin E. A social-ecologic approach to assessing support for disease self-management: the Chronic Illness Resources Survey. J Behav Med. 2000 Dec;23(6):559-83. doi: 10.1023/a:1005507603901. PMID 11199088
- [Background] Glasgow RE, Toobert DJ, Barrera M Jr, Strycker LA. The Chronic Illness Resources Survey: cross-validation and sensitivity to intervention. Health Educ Res. 2005 Aug;20(4):402-9. doi: 10.1093/her/cyg140. Epub 2004 Nov 30. PMID 15572438
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] Haaxma CA, Bloem BR, Borm GF, Oyen WJ, Leenders KL, Eshuis S, Booij J, Dluzen DE, Horstink MW. Gender differences in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2007 Aug;78(8):819-24. doi: 10.1136/jnnp.2006.103788. Epub 2006 Nov 10. PMID 17098842
- [Background] Habermann B. Continuity challenges of Parkinson's disease in middle life. J Neurosci Nurs. 1999 Aug;31(4):200-7. doi: 10.1097/01376517-199908000-00001. PMID 10553567
- [Background] Habermann B, Davis LL. Caring for family with Alzheimer's disease and Parkinson's disease: needs, challenges and satisfaction. J Gerontol Nurs. 2005 Jun;31(6):49-54. doi: 10.3928/0098-9134-20050601-11. PMID 16138530
- [Background] Harezlak J, Naumova E, Laird NM. LongCriSP: a test for bump hunting in longitudinal data. Stat Med. 2007 Mar 15;26(6):1383-97. doi: 10.1002/sim.2623. PMID 16850452
- [Background] Hemmesch AR, Tickle-Degnen L, Zebrowitz LA. The influence of facial masking and sex on older adults' impressions of individuals with Parkinson's disease. Psychol Aging. 2009 Sep;24(3):542-9. doi: 10.1037/a0016105. PMID 19739910
- [Background] Holman HR, Lorig KR. Overcoming barriers to successful aging. Self-management of osteoarthritis. West J Med. 1997 Oct;167(4):265-8. No abstract available. PMID 9348758
- [Background] Holt-Lunstad J, Smith TB, Layton JB. Social relationships and mortality risk: a meta-analytic review. PLoS Med. 2010 Jul 27;7(7):e1000316. doi: 10.1371/journal.pmed.1000316. PMID 20668659
- [Background] Horton NJ, Laird NM, Murphy JM, Monson RR, Sobol AM, Leighton AH. Multiple informants: mortality associated with psychiatric disorders in the Stirling County Study. Am J Epidemiol. 2001 Oct 1;154(7):649-56. doi: 10.1093/aje/154.7.649. PMID 11581099
- [Background] Hunt SM, McEwen J. The development of a subjective health indicator. Sociol Health Illn. 1980 Nov;2(3):231-46. doi: 10.1111/1467-9566.ep11340686. No abstract available. PMID 10298135
- [Background] Karlsen KH, Tandberg E, Arsland D, Larsen JP. Health related quality of life in Parkinson's disease: a prospective longitudinal study. J Neurol Neurosurg Psychiatry. 2000 Nov;69(5):584-9. doi: 10.1136/jnnp.69.5.584. PMID 11032608
- [Background] Litwin H. Social networks and well-being: a comparison of older people in Mediterranean and non-Mediterranean countries. J Gerontol B Psychol Sci Soc Sci. 2010 Sep;65(5):599-608. doi: 10.1093/geronb/gbp104. Epub 2009 Dec 14. PMID 20008485
- [Background] Lyons KD, Hull JG, Root LD, Kimtis E, Schaal AD, Stearns DM, Williams IC, Meehan KR, Ahles TA. A pilot study of activity engagement in the first six months after stem cell transplantation. Oncol Nurs Forum. 2011 Jan;38(1):75-83. doi: 10.1188/11.ONF.75-83. PMID 21186163
- [Background] Lyons KD, Tickle-Degnen L. Reliability and validity of a videotape method to describe expressive behavior in persons with Parkinson's disease. Am J Occup Ther. 2005 Jan-Feb;59(1):41-9. doi: 10.5014/ajot.59.1.41. PMID 15707122
- [Background] Martinez LS, Rubin CL, Russell B, Leslie LK, Brugge D. Community conceptualizations of health: implications for transdisciplinary team science. Clin Transl Sci. 2011 Jun;4(3):163-7. doi: 10.1111/j.1752-8062.2011.00289.x. PMID 21707945
- [Background] Martinez-Martin P, Forjaz MJ, Frades-Payo B, Rusinol AB, Fernandez-Garcia JM, Benito-Leon J, Arillo VC, Barbera MA, Sordo MP, Catalan MJ. Caregiver burden in Parkinson's disease. Mov Disord. 2007 May 15;22(7):924-31; quiz 1060. doi: 10.1002/mds.21355. PMID 17238193
- [Background] McRae C, Fazio E, Hartsock G, Kelley L, Urbanski S, Russell D. Predictors of loneliness in caregivers of persons with Parkinson's disease. Parkinsonism Relat Disord. 2009 Sep;15(8):554-7. doi: 10.1016/j.parkreldis.2009.01.007. Epub 2009 Feb 28. PMID 19251464
- [Background] Naumova EN, Must A, Laird NM. Tutorial in Biostatistics: Evaluating the impact of 'critical periods' in longitudinal studies of growth using piecewise mixed effects models. Int J Epidemiol. 2001 Dec;30(6):1332-41. doi: 10.1093/ije/30.6.1332. PMID 11821342
- [Background] Nazem S, Siderowf AD, Duda JE, Have TT, Colcher A, Horn SS, Moberg PJ, Wilkinson JR, Hurtig HI, Stern MB, Weintraub D. Montreal cognitive assessment performance in patients with Parkinson's disease with "normal" global cognition according to mini-mental state examination score. J Am Geriatr Soc. 2009 Feb;57(2):304-8. doi: 10.1111/j.1532-5415.2008.02096.x. Epub 2008 Dec 10. PMID 19170786
- [Background] Netuveli G, Wiggins RD, Montgomery SM, Hildon Z, Blane D. Mental health and resilience at older ages: bouncing back after adversity in the British Household Panel Survey. J Epidemiol Community Health. 2008 Nov;62(11):987-91. doi: 10.1136/jech.2007.069138. PMID 18854503
- [Background] Nolte S, Elsworth GR, Sinclair AJ, Osborne RH. The extent and breadth of benefits from participating in chronic disease self-management courses: a national patient-reported outcomes survey. Patient Educ Couns. 2007 Mar;65(3):351-60. doi: 10.1016/j.pec.2006.08.016. Epub 2006 Oct 5. PMID 17027221
- [Background] Peto V, Jenkinson C, Fitzpatrick R. PDQ-39: a review of the development, validation and application of a Parkinson's disease quality of life questionnaire and its associated measures. J Neurol. 1998 May;245 Suppl 1:S10-4. doi: 10.1007/pl00007730. PMID 9617716
- [Background] Pinquart M, Sorensen S. Influences of socioeconomic status, social network, and competence on subjective well-being in later life: a meta-analysis. Psychol Aging. 2000 Jun;15(2):187-224. doi: 10.1037//0882-7974.15.2.187. PMID 10879576
- [Background] Post B, Muslimovic D, van Geloven N, Speelman JD, Schmand B, de Haan RJ; CARPA-study group. Progression and prognostic factors of motor impairment, disability and quality of life in newly diagnosed Parkinson's disease. Mov Disord. 2011 Feb 15;26(3):449-56. doi: 10.1002/mds.23467. Epub 2011 Feb 10. PMID 21312273
- [Background] Rao D, Choi SW, Victorson D, Bode R, Peterman A, Heinemann A, Cella D. Measuring stigma across neurological conditions: the development of the stigma scale for chronic illness (SSCI). Qual Life Res. 2009 Jun;18(5):585-95. doi: 10.1007/s11136-009-9475-1. Epub 2009 Apr 25. PMID 19396572
- [Background] Reuther M, Spottke EA, Klotsche J, Riedel O, Peter H, Berger K, Athen O, Kohne-Volland R, Dodel RC. Assessing health-related quality of life in patients with Parkinson's disease in a prospective longitudinal study. Parkinsonism Relat Disord. 2007 Mar;13(2):108-14. doi: 10.1016/j.parkreldis.2006.07.009. Epub 2006 Oct 19. PMID 17055326
- [Background] Roger KS, Medved MI. Living with Parkinson's disease-managing identity together. Int J Qual Stud Health Well-being. 2010 Mar 30;5(2). doi: 10.3402/qhw.v5i2.5129. PMID 20640016
- [Background] Sarkar R, Ajjampur SS, Ward HD, Kang G, Naumova EN. Analysis of human immune responses in quasi-experimental settings: tutorial in biostatistics. BMC Med Res Methodol. 2012 Jan 3;12:1. doi: 10.1186/1471-2288-12-1. PMID 22214542
- [Background] Schulman EA, Hohler AD. The American Academy of Neurology position statement on abuse and violence. Neurology. 2012 Feb 7;78(6):433-5. doi: 10.1212/WNL.0b013e318245d21c. Epub 2012 Jan 25. No abstract available. PMID 22282648
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Skodda S, Rinsche H, Schlegel U. Progression of dysprosody in Parkinson's disease over time--a longitudinal study. Mov Disord. 2009 Apr 15;24(5):716-22. doi: 10.1002/mds.22430. PMID 19117364
- [Background] Stokols D, Grzywacz JG, McMahan S, Phillips K. Increasing the health promotive capacity of human environments. Am J Health Promot. 2003 Sep-Oct;18(1):4-13. doi: 10.4278/0890-1171-18.1.4. PMID 13677958
- [Background] Sunvisson H, Habermann B, Weiss S, Benner P. Augmenting the Cartesian medical discourse with an understanding of the person's lifeworld, lived body, life story and social identity. Nurs Philos. 2009 Oct;10(4):241-52. doi: 10.1111/j.1466-769X.2009.00413.x. PMID 19743968
- [Background] Takahashi K, Tickle-Degnen L, Coster WJ, Latham NK. Expressive behavior in Parkinson's disease as a function of interview context. Am J Occup Ther. 2010 May-Jun;64(3):484-95. doi: 10.5014/ajot.2010.09078. PMID 20608279
- [Background] Tanji H, Anderson KE, Gruber-Baldini AL, Fishman PS, Reich SG, Weiner WJ, Shulman LM. Mutuality of the marital relationship in Parkinson's disease. Mov Disord. 2008 Oct 15;23(13):1843-9. doi: 10.1002/mds.22089. PMID 18759355
- [Background] Tickle-Degnen L, Ellis T, Saint-Hilaire MH, Thomas CA, Wagenaar RC. Self-management rehabilitation and health-related quality of life in Parkinson's disease: a randomized controlled trial. Mov Disord. 2010 Jan 30;25(2):194-204. doi: 10.1002/mds.22940. PMID 20077478
- [Background] Tickle-Degnen L, Lyons KD. Practitioners' impressions of patients with Parkinson's disease: the social ecology of the expressive mask. Soc Sci Med. 2004 Feb;58(3):603-14. doi: 10.1016/s0277-9536(03)00213-2. PMID 14652056
- [Background] Tickle-Degnen L, Zebrowitz LA, Ma HI. Culture, gender and health care stigma: Practitioners' response to facial masking experienced by people with Parkinson's disease. Soc Sci Med. 2011 Jul;73(1):95-102. doi: 10.1016/j.socscimed.2011.05.008. Epub 2011 May 25. PMID 21664737
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Wright Willis A, Evanoff BA, Lian M, Criswell SR, Racette BA. Geographic and ethnic variation in Parkinson disease: a population-based study of US Medicare beneficiaries. Neuroepidemiology. 2010;34(3):143-51. doi: 10.1159/000275491. Epub 2010 Jan 15. PMID 20090375
- [Background] Willis AW, Schootman M, Evanoff BA, Perlmutter JS, Racette BA. Neurologist care in Parkinson disease: a utilization, outcomes, and survival study. Neurology. 2011 Aug 30;77(9):851-7. doi: 10.1212/WNL.0b013e31822c9123. Epub 2011 Aug 10. PMID 21832214
- [Background] Worth A, Tierney AJ. Conducting research interviews with elderly people by telephone. J Adv Nurs. 1993 Jul;18(7):1077-84. doi: 10.1046/j.1365-2648.1993.18071077.x. PMID 8370897
- [Background] Jenkinson C., Fitzpatrick R., Peto V., Greenhall R. and Hyman N. (1997). The PDQ-8: Development and validation of a short-form Parkinson"s disease questionnaire. Psychology and Health, 12, 805-814.
- [Background] Baum, C.M., & Edwards, D. (2008). Activity Card Sort, 2nd ed., AOTA Press, Bethesda, MD.
- [Background] Pennebaker, J. W., Booth, R. J. & Francis, M. E., & (2007). Linguistic Inquiry and Word Count (LIWC). [Computer software]. Austin, TX: LIWC.net.
- [Background] Sheikh, J., & Yesavage, J. (1986). Geriatric Depression Scale (GDS): Recent evidence and development of a shorter version. In T.L. Brink (Ed.), Clinical Gerontology: A guide to assessment and intervention (pp. 165-173). New York: Haworth Press.
- [Background] Svestkova O. International classification of functioning, disability and health of World Health Organization (ICF). Prague Med Rep. 2008;109(4):268-74. PMID 19537677
- [Result] Sprague Martinez L, Thomas CA, Saint-Hilaire M, McLaren J, Young J, Habermann B, Tickle-Degnen L. Using a Macro Social Work Strategy to Improve Outreach in Parkinson's Disease Research. Soc Work. 2018 Jul 1;63(3):265-268. doi: 10.1093/sw/swy026. No abstract available. PMID 29722873
- [Result] Berger S, Chen T, Eldridge J, Thomas CA, Habermann B, Tickle-Degnen L. The self-management balancing act of spousal care partners in the case of Parkinson's disease. Disabil Rehabil. 2019 Apr;41(8):887-895. doi: 10.1080/09638288.2017.1413427. Epub 2017 Dec 12. PMID 29228835
- [Result] Gunnery SD, Naumova EN, Saint-Hilaire M, Tickle-Degnen L. Mapping spontaneous facial expression in people with Parkinson's disease: A multiple case study design. Cogent Psychol. 2017;4:1376425. doi: 10.1080/23311908.2017.1376425. Epub 2017 Sep 8. PMID 29607351
- [Result] Gunnery SD, Habermann B, Saint-Hilaire M, Thomas CA, Tickle-Degnen L. The Relationship between the Experience of Hypomimia and Social Wellbeing in People with Parkinson's Disease and their Care Partners. J Parkinsons Dis. 2016 Jun 3;6(3):625-30. doi: 10.3233/JPD-160782. PMID 27285568
- [Result] Ma HI, Saint-Hilaire M, Thomas CA, Tickle-Degnen L. Stigma as a key determinant of health-related quality of life in Parkinson's disease. Qual Life Res. 2016 Dec;25(12):3037-3045. doi: 10.1007/s11136-016-1329-z. Epub 2016 Jun 3. PMID 27259581
- [Result] Tickle-Degnen L, Saint-Hilaire M, Thomas CA, Habermann B, Martinez LS, Terrin N, Noubary F, Naumova EN. Emergence and evolution of social self-management of Parkinson's disease: study protocol for a 3-year prospective cohort study. BMC Neurol. 2014 May 2;14:95. doi: 10.1186/1471-2377-14-95. PMID 24885181

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT03938974/Prot_SAP_000.pdf